CLINICAL TRIAL: NCT06768086
Title: 3 Months Preoperative Administration of Eutris Plus Prior Hysteroscopic Myomectomy: a Pilot Study
Brief Title: Preoperative Administration of EGCG, Vitamin D and DCI Prior Hysteroscopic Myomectomy
Acronym: PREHYSMYOM
Status: Completed | Type: Observational
Sponsor: Centro di Ricerca Clinica Salentino (Network)
Responsible Party: Sponsor
Other Study IDs: CER1024
Record Dates: First submitted 2024-12-31; First posted 2025-01-10 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2024-12

CONDITIONS: Uterine Fibroids; Hysteroscopic Myomectomy; Treatment Compliance; Patient Compliance; Treatment Complication
Keywords: uterine fibroid; uterine myoma; hysteroscopic myomectomy; D-Chiro-Inositol; Epigallocatechin Gallate; Vitamin D; Surgical complication
MeSH Terms: conditions — Leiomyoma; Patient Compliance; Myofibroma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treated patiens' Group as Group 1: Pre-treated patients by Eutris Plus for 3 months and the hysteroscopic myomectomy
  Interventions: Procedure: Hysteroscopic myomectomy
- Untreated patiens' Group as Group 2: Control group of women (no treatments and without preoperative hormonal therapy) scheduled to undergo hysteroscopic myomectomy after 3 months.
  Interventions: Procedure: Hysteroscopic myomectomy

INTERVENTIONS:
Procedure: Hysteroscopic myomectomy — The hysteroscopic myomectomies were conducted during the follicular phase of the menstrual cycle. Throughout the surgical procedure, the intrauterine pressure was meticulously maintained at less than 80 mm Hg. Data on the duration of the surgical intervention, the volume of fluid administered, and the volume of fluid absorbed were collected. Complete resection was characterized as the total excision of the myoma. The determination of the completeness of myomectomy was made by the experienced surgeon during the surgical process. In instances where the resection was deemed incomplete, the decision to pursue a secondary surgical intervention was predicated on ultrasonographic evaluations, the symptomatic presentation of the patients, and, in certain circumstances, the findings from diagnostic hysteroscopy. Cases in which access to the uterine cavity was unfeasible were classified as "failed procedures" and were subsequently excluded from the study.

SUMMARY:
The administration of Epigallocatechin gallate (EGCG), Vitamin D and D-Chiro-Inositol (DCI) are effective in reducing the volume of fibroids and improving the symptoms of uterine fibroids.

Since this benefit has been seen in laparoscopic myomectomy, a study was designed to see if there are positive effects in women undergoing hysteroscopic myomectomy.

For this reason, patients were enrolled to undergo hysteroscopic myomectomy, then divided into two groups: patients to be treated preoperatively with a product based on Epigallocatechin gallate (EGCG), Vitamin D and D-Chiro-Inositol (DCI) for 3 months before myomectomy and patients not to be treated before surgery. All clinical and surgical parameters were then collected and analyzed to verify the differences between the two groups (treated women VS untreated women).

DETAILED DESCRIPTION:
The administration of Epigallocatechin gallate (EGCG), Vitamin D and D-Chiro-Inositol (DCI) are effective in reducing the volume of fibroids and improving the symptoms of uterine fibroids.

Since this benefit has been seen in laparoscopic myomectomy, a study was designed to see if there are positive effects in women undergoing hysteroscopic myomectomy.

For this reason, patients were enrolled to undergo hysteroscopic myomectomy, then divided into two groups: patients to be treated preoperatively with a product based on Epigallocatechin gallate (EGCG), Vitamin D and D-Chiro-Inositol (DCI) for 3 months before myomectomy and patients not to be treated before surgery.

The ideal objectives of a preoperative treatment in patients undergoing hysteroscopic myomectomy are to facilitate surgery (i.e, better visualization of the uterine cavity, decrease in the length of the procedure), to improve the characteristics of myomas (such as decreasing their volume and vascularization) and of endometrium (inducing endometrial atrophy and ideally amenorrhea, that can be useful for scheduling surgery and recovering from anemia), and to decrease the risk of intraoperative complications (such as uterine perforation, excessive bleeding, and fluid intravasation), the rate of 2-step hysteroscopic procedures, and ideally, the risk of long-term complications (such as intrauterine adhesions).

Generally, the main disadvantages of preoperative medications are treatment-related adverse effects, cost, and delay in surgery.

Since these are natural molecules, all contained in a commonly sold supplement (EUTRIS PLUS), many patients have willingly agreed to take it for 3 months before surgery.

Thus, the aim of the study was if the Eutris Plus administration can facilitate hysteroscopic myomectomy by decreasing myoma volume and vascularization, even not inducing endometrial atrophy.

Study setting: Prospective, observational study on type of Submucous Myomas to be resected (FIGO type 0, 1, 2), by bipolar hysteroscopic resectoscopy (with use of bipolar saline solutions), performed from the fifth to the 15th day after the end of the menstrual cycle.

Informed consent was obtained from all individual participants included in the study.

Patients' settings in the two arms:

1. Pre-treated patients by Eutris Plus for 3 months and the hysteroscopic myomectomy.
2. Control group of women (no treatments and without preoperative hormonal therapy) scheduled to undergo hysteroscopic myomectomy after 3 months.

Therapy by a total of 300 mg EGCG, 50 μg vitamin D, and 50 mg DCI divided in 2 pills per day for 3 months.

Patients were informed that Eutris Plus decreases uterine myoma volume and improves iron-deficiency anemia.

However, they were also informed that limited data are available on the usefulness of Eutris Plus before hysteroscopic resection under general anesthesia and that no previous study investigated the role of Eutris Plus before hysteroscopic myomectomy.

The hysteroscopies were conducted during the follicular phase of the menstrual cycle in participants who did not undergo preoperative intervention and during the interval after the conclusion of Eutris Plus treatment and preceding the initial menstrual cycle in individuals receiving preoperative therapy.

Throughout the hysteroscopic myomectomy, the intrauterine pressure was meticulously maintained at less than 80 mm Hg.

The duration of the surgical intervention, the volume of fluid administered, and the volume of fluid absorbed were systematically documented.

Complete resection was characterized as the total excision of the myoma; however, it was acknowledged that certain fragments of the myoma remained within the uterine cavity. The determination of the completeness of myomectomy was made by the experienced surgeon during the surgical process.

In instances where the resection was deemed incomplete, the decision to pursue a secondary surgical intervention was predicated on ultrasonographic evaluations, the symptomatic presentation of the patients, and, in certain circumstances, the findings from diagnostic hysteroscopy.

Cases in which access to the uterine cavity was unfeasible were classified as "failed procedures" and were subsequently excluded from the study.

At the conclusion of each surgical intervention, the surgeon was obliged to complete a form evaluating the surgical experience, which was based on six specific items with corresponding scoring metrics.

In hysteroscopic myomectomies, the overall surgical experience score was: the sum of the visualization, myoma-myometrium delineation, extrusion, fluid deficit, blood loss, and overall ease of treatment scores, thus surgeons evaluated:

1. hysteroscopic visualization (excellent [score = 3]; good [2]; or satisfactory, poor, or very poor [1])
2. relationship to the myometrium (well delineated [3]; well delineated in some areas, poor in others [2]; or poorly delineated throughout [1])
3. extrusion into the cavity during the procedure (yes [2] or no [1])
4. distension fluid deficit (<250 mL [3], 250-500 mL [2], or >500 mL [1])
5. estimated blood loss (<50 mL [3], 50-100 mL [2] or >100 mL [1])
6. overall ease of the procedure compared with other similar cases (easier [3], routine [2], or more difficult [1]) The overall hysteroscopic surgical experience score was determined by summing the scores for each subscale for a total of 6 to 17, with higher scores indicating a better surgical experience.

Surgeons were blinded to the eventual preoperative treatment (the decision whether or not to take the therapy was made in the outpatient clinic at the time of enrollment), so their experiences have been wide from any preconceived beliefs about medical pretreatment.

Main short term-Outcomes items were:

1. Patients' characteristics
2. Change in myoma volume by Eutris Plus after 3 months
3. Surgical parameters
4. Complete/incomplete myoma resection
5. Surgical complications
6. Patients' satisfaction (at Hospital dismissal, generally in the late afternoon, after almost 5 hours) The Patients did perceive, before hospital discharge, the global operative procedure using a 10-point visual analog scale (VAS), to be filled out and inserted into the medical record.

The primary objective of the study was to compare the operative results between the 2 study groups: duration of surgery, the volume of fluid infused, and the volume of fluid absorbed.

The secondary objective of the study was to compare the rate of complete resections in the 2 study groups.

The tertiary objective of the study was to assess the surgical complications and patients' compliance in patients treated with Eutris plus.

According to literature evidence - and our clinical experience - hysteroscopic myomectomy requires on average 45 to 60 minutes per surgical intervention. Considering our surgical report, we estimated an expected average of 55 ± 15 minutes per surgical procedure. Setting an anticipated results of 45 minutes per surgery in the intervention group and choosing an alpha equal to 0.05 and a power equal to 85%, we calculated 40 patients per group. Considering a potential dropout equal to 20%, we decided to enroll 48 patients per arm.

Comparative analyses of categorical data were executed utilizing the Fisher exact test, whereas analyses of continuous data were performed using the Student-t test.

All statistical evaluations were conducted utilizing SAS (Version 9.3; SAS Institute, Cary, NC).

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of FIGO type 0 to 2 fibroids, with a diameter of 20 - 35 mm. Must be able to swallow tablets.

Exclusion Criteria:

Clinical diagnosis of polyps associated to FIGO type 0 to 2 fibroids. Non-hysteroscopic surgical procedures. The presence of more than 2 FIGO type 0 to 2 fibroids.

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women
Study Population: Women of reproductive age, in good health, without pathologies compromising general anesthesia and willing to participate in the study, on a voluntary basis.
  The decision about whether to pretreat patients medically or not, was twice:
  1. patient' preference design.
  2. if the patients were undecided, at the discretion of the staff physician, as was the choice of therapy.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Operative results | 8 months
  to compare the operative results between the 2 study groups: duration of surgery in min
Surgical results | 8 months
  to compare the operative results between the 2 study groups: the volume of fluid infused in ml
Hysteroscopic results | 8 months
  to compare the operative results between the 2 study groups: the volume of fluid absorbed in ml

SECONDARY OUTCOMES:
Complete resection of fibroids | 8 months
  to compare the rate of complete fibroids' resections in the 2 study groups.

OTHER OUTCOMES:
Patients' complications | 8 months
  to assess the percentage of surgical complications in patients treated with Eutris plus.
Patients' compliance | 8 months
  to assess the percentage of patients' positive compliance in patients treated with Eutris plus.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Tinelli, MD, Principal Investigator — Veris delli Ponti Hospital Scorrano, 73020 Lecce, Italy
Locations (1):
- Ospedale Veris delli Ponti, Scorrano, Lecce, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tinelli A, Gustapane S, D'Oria O, Licchelli M, Panese G. Nutraceuticals in fibroid management after ulipristal acetate administration: An observational study on patients' compliance. Int J Gynaecol Obstet. 2022 Jan;156(1):133-138. doi: 10.1002/ijgo.13692. Epub 2021 May 5. PMID 33797759
- [Result] Tinelli A, Panese G, Licchelli M, Morciano A, Pecorella G, Gambioli R. The impact of epigallocatechin gallate, vitamin D, and D-chiro-inositol on early surgical outcomes of laparoscopic myomectomy: a pilot study. Arch Gynecol Obstet. 2024 Mar;309(3):1021-1026. doi: 10.1007/s00404-023-07324-x. Epub 2024 Jan 6. PMID 38183422
- [Result] Vafaei S, Ciebiera M, Omran MM, Ghasroldasht MM, Yang Q, Leake T, Wolfe R, Ali M, Al-Hendy A. Evidence-Based Approach for Secondary Prevention of Uterine Fibroids (The ESCAPE Approach). Int J Mol Sci. 2023 Nov 4;24(21):15972. doi: 10.3390/ijms242115972. PMID 37958957
- [Result] Ali M, Ciebiera M, Wlodarczyk M, Alkhrait S, Maajid E, Yang Q, Hsia SM, Al-Hendy A. Current and Emerging Treatment Options for Uterine Fibroids. Drugs. 2023 Dec;83(18):1649-1675. doi: 10.1007/s40265-023-01958-6. Epub 2023 Nov 3. PMID 37922098
- [Result] Lethaby A, Puscasiu L, Vollenhoven B. Preoperative medical therapy before surgery for uterine fibroids. Cochrane Database Syst Rev. 2017 Nov 15;11(11):CD000547. doi: 10.1002/14651858.CD000547.pub2. PMID 29139105
- [Result] Wlodarczyk M, Ciebiera M, Nowicka G, Lozinski T, Ali M, Al-Hendy A. Epigallocatechin Gallate for the Treatment of Benign and Malignant Gynecological Diseases-Focus on Epigenetic Mechanisms. Nutrients. 2024 Feb 17;16(4):559. doi: 10.3390/nu16040559. PMID 38398883
- [Result] Kamal DAM, Salamt N, Zaid SSM, Mokhtar MH. Beneficial Effects of Green Tea Catechins on Female Reproductive Disorders: A Review. Molecules. 2021 May 3;26(9):2675. doi: 10.3390/molecules26092675. PMID 34063635
- [Result] Hazimeh D, Massoud G, Parish M, Singh B, Segars J, Islam MS. Green Tea and Benign Gynecologic Disorders: A New Trick for An Old Beverage? Nutrients. 2023 Mar 16;15(6):1439. doi: 10.3390/nu15061439. PMID 36986169
- [Result] Krzyzanowski J, Paszkowski T, Wozniak S. The Role of Nutrition in Pathogenesis of Uterine Fibroids. Nutrients. 2023 Dec 1;15(23):4984. doi: 10.3390/nu15234984. PMID 38068842
- [Result] Szydlowska I, Nawrocka-Rutkowska J, Brodowska A, Marciniak A, Starczewski A, Szczuko M. Dietary Natural Compounds and Vitamins as Potential Cofactors in Uterine Fibroids Growth and Development. Nutrients. 2022 Feb 9;14(4):734. doi: 10.3390/nu14040734. PMID 35215384
- [Result] Arjeh S, Darsareh F, Asl ZA, Azizi Kutenaei M. Effect of oral consumption of vitamin D on uterine fibroids: A randomized clinical trial. Complement Ther Clin Pract. 2020 May;39:101159. doi: 10.1016/j.ctcp.2020.101159. Epub 2020 Apr 2. PMID 32379687
- [Result] Combs A, Singh B, Nylander E, Islam MS, Nguyen HV, Parra E, Bello A, Segars J. A Systematic Review of Vitamin D and Fibroids: Pathophysiology, Prevention, and Treatment. Reprod Sci. 2023 Apr;30(4):1049-1064. doi: 10.1007/s43032-022-01011-z. Epub 2022 Aug 12. PMID 35960442
- [Result] Vergara D, Catherino WH, Trojano G, Tinelli A. Vitamin D: Mechanism of Action and Biological Effects in Uterine Fibroids. Nutrients. 2021 Feb 11;13(2):597. doi: 10.3390/nu13020597. PMID 33670322
- [Result] Porcaro G, Santamaria A, Giordano D, Angelozzi P. Vitamin D plus epigallocatechin gallate: a novel promising approach for uterine myomas. Eur Rev Med Pharmacol Sci. 2020 Mar;24(6):3344-3351. doi: 10.26355/eurrev_202003_20702. PMID 32271452
- [Result] Grandi G, Del Savio MC, Melotti C, Feliciello L, Facchinetti F. Vitamin D and green tea extracts for the treatment of uterine fibroids in late reproductive life: a pilot, prospective, daily-diary based study. Gynecol Endocrinol. 2022 Jan;38(1):63-67. doi: 10.1080/09513590.2021.1991909. Epub 2021 Oct 16. PMID 34658291